CLINICAL TRIAL: NCT05005715
Title: Effect of Dexmedetomidine on Intraoperative Neuroendocrine Stress Response and Early Postoperative Quality of Recovery in Non-functioning Pituitary Adenoma Patients Undergoing Endoscopic Transsphenoidal Tumor Surgery
Brief Title: Effect of Dexmedetomidine on Quality of Recovery in Non-functioning Pituitary Adenoma Patients Undergoing Endoscopic Transsphenoidal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TSA_precedex
Record Dates: First submitted 2021-07-26; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Non-functioning Pituitary Adenoma
Keywords: non-functioning Pituitary Adenoma; endoscopic transsphenoidal tumor surgery; dexmedetomidine; quality of recovery
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator): After the induction of anesthesia, the dexmedetomidine group received intravenous dexmedetomidine at a loading dose of 1µg/kg for 10 min, followed by a maintenance dose of 0.5µg/kg/h until the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): After the induction of anesthesia, the control group received intravenous normal saline at the same loading volume for 10 min, followed by the same volume until the end of surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients were randomly assigned to the dexmedetomidine or control group. Dexmedetomidine group received intravenous dexmedetomidine and control group received intravenous normal saline during surgery.
  Arms: Dexmedetomidine group
Drug: normal saline — Patients were randomly assigned to the dexmedetomidine or control group. Dexmedetomidine group received intravenous dexmedetomidine and control group received intravenous normal saline during surgery.
  Arms: Control group

SUMMARY:
In multiple previous studies that have explored the use of dexmedetomidine in transsphenoidal tumor resection surgery, dexmedetomidine showed many beneficial effects like reducing the requirement of analgesics and anesthetics, improving hemodynamic stability and decreasing the emergence time, extubation time and visual analog scale at emergence. Therefore, the investigators hypothesized that dexmedetomidine would decrease neuroendocrine stress response and improve the quality of postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Non-functioning patients undergoing endoscopic transsphenoidal tumor surgery under general anesthesia

Exclusion Criteria:

* Patients who do not agree to participate in the study
* Patients with contraindication to dexmedetomidine
* Patients with previous history of endoscopic transsphenoidal tumor surgery
* Patients who take anticoagulants or have bleeding disorder
* Patients with conduction block or cardiovascular disease
* Patients with psychiatric disease such as dementia, delirium
* Patients have difficulty filling out the QoR-15 questionnaire
* Pregnant or lactating women
* Patients who have allergies to propofol, remifentanil, fentanyl or rocuronium
* Patients with myasthenia gravis or myasthenic syndrome

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2022-08-29 (Estimated); Study Completion 2023-08-29 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery-15 (QoR-15) score | postoperative day 1
  Self-rated questionnaire composed of 15 items (each item: 0-10 points, total: 0-150 points) of five dimensions: physical well-being, physical independence, emotional state, psychological support, and pain. Higher scores indicate better quality of recovery.

SECONDARY OUTCOMES:
Serum level of triiodothyronine (T3) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ng/dL
Serum level of triiodothyronine (T4) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ng/dL
Serum level of thyroid stimulating hormone (TSH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  uIU/mL
Serum level of luteinizing hormone (LH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  mIU/mL
Serum level of follicle stimulating hormone (FSH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  mIU/mL
Serum level of adredocorticotrophic hormone (ACTH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  pg/mL
Serum level of growth hormone (GH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ng/mL
Serum level of insulin-like growth factor-1 (IGF-1) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ng/mL
Serum level of prolactin | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ng/mL
Serum level of antidiuretic hormone (ADH) | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  pg/ml
Serum level of cortisol | preoperative (1-2 month before surgery), intraoperative (when surgeon starts tumor resection), immediately postoperative (30 min after the end of surgery)
  ug/dL
Pain score (visual analogue scale, VAS) | postoperative 4 hour, 1 day, 2 day
  Self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Time to the first administration of rescue analgesics after the end of surgery | postoperative (up to 2 weeks after surgery)
Total amounts of rescue analgesics | postoperative (up to 2 weeks after surgery)
Total amounts of propofol and remifentanil administered during surgery | intraoperative (from induction of anesthesia until end of anesthesia)
Time to emergence after the end of surgery | postoperative (up to 1 day after surgery)
Time to extubation after the end of surgery | postoperative (up to 1 day after surgery)
Incidence and severity of postoperative complications | postoperative (up to 2 weeks after surgery)
  nausea, vomiting, etc.
Hospital length of stay | postoperative (up to 2 weeks after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No